CLINICAL TRIAL: NCT04212819
Title: Comparison of Oxidative Stress and Asymmetric Dimethyl Arginine Levels Before and After Erythrocyte Suspension Transfusion
Brief Title: Before and After Erythrocyte Suspension Transfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Erhan BOZKURT, Assistant Professor, Afyonkarahisar Health Sciences University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2015/7-165
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Anemia; Oxidative Stress
Keywords: Erythrocyte suspension; Total antioxidant status; Total oxidant status; Asymmetric dimethylarginine
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before erythrocyte suspension (ES) transfusion group (Experimental): 50 (Female/Male: 25/25) patients were included in this study. Total antioxidant status (TAS), total oxidant status (TOS) and ADMA levels were measured from the patients after diagnoses of anemia.
  Interventions: Other: Before Erythrocyte Suspension (ES)
- After erythrocyte suspension transfusion group (Experimental): 24 hours after ES transfusion, total antioxidant status (TAS), total oxidant status (TOS) and ADMA levels were measured from the patients.
  Interventions: Other: After Erythrocyte Suspension (ES)

INTERVENTIONS:
Other: Before Erythrocyte Suspension (ES) — ES transfusion needs of the patients were determined according to clinical signs and symptoms. Vital signs were closely monitored and recorded before, during and after transfusion. Infusion was performed slowly for the first 15 minutes in terms of allergic reaction, and then the transfusion rate was adjusted according to the patient's clinic.
  Arms: Before erythrocyte suspension (ES) transfusion group
Other: After Erythrocyte Suspension (ES) — Venous blood samples were obtained from patients who needed ES transfusion before transfusion. Control venous blood samples were obtained from the patients who did not develop any complications for 24 hours after starting of the transfusion and became hemodynamically stable.
  Arms: After erythrocyte suspension transfusion group

SUMMARY:
Hypoperfusion, hypoxia and ischemia occurs in circulation as a result of anemia. All of these situations lead to oxidative stress and endothelial dysfunction in the organism. In this study, the investigators aimed to investigate the oxidant-antioxidant balance and asymmetric dimethylarginine (ADMA) levels in patients that have symptomatic anemia in need of erythrocyte suspension (ES) transfusion. To the best of the investigators knowledge, there have been few studies in the literature on anemia and total oxidant, total antioxidant and ADMA levels. We aimed to observe changes in oxidative - antioxidant ADMA levels before and after ES transfusion.

ELIGIBILITY:
Inclusion Criteria:

* Only patients with deep anemia and anemia due to gastrointestinal bleeding patients in need of erythrocyte suspension transfusion were included.

Exclusion Criteria:

* Patients with history of hypertension, diabetes, coronary artery disease, congestive heart failure, chronic renal failure, liver failure were not included to the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-04-01 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Whole Blood Count Test | 24 hour
  Patients with deep anemia and anemia due to gastrointestinal bleeding patients in need of erythrocyte suspension transfusion were included. ES transfusion needs of the patients were determined according to clinical signs and symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan BOZKURT, M.D., Principal Investigator — Afyonkarahisar Health Sciences University